CLINICAL TRIAL: NCT02498639
Title: Comparison of Safety and Efficacy of Percutaneous Balloon Aortic Valvuloplasty Performed With or Without Rapid Ventricular Pacing - The Pacing vs No Pacing Study (PNP Study)
Brief Title: The Pacing vs No Pacing Study - PNP Study
Acronym: PNP
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Dr. Antonio Marzocchi, MD, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CE41/2015/O/Sper
Record Dates: First submitted 2015-07-10; First posted 2015-07-15 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-07

CONDITIONS: Aortic Valve Stenosis
Keywords: balloon aortic valvuloplasty; rapid ventricular pacing; outcome
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BAV without pacing (Active Comparator): Patients undergo percutaneous balloon aortic valvuloplasty (BAV) without previous insertion of a temporary pacemaker lead in the right ventricle. Stabilization of the balloon during inflation is done without rapid pacing.
  Interventions: Procedure: percutaneous balloon aortic valvuloplasty
- BAV with pacing (Active Comparator): Patients undergo percutaneous balloon aortic valvuloplasty (BAV) after previous insertion of a temporary pacemaker lead in the right ventricle. Stabilization of the balloon during inflation is done under rapid pacing.
  Interventions: Procedure: percutaneous balloon aortic valvuloplasty

INTERVENTIONS:
Procedure: percutaneous balloon aortic valvuloplasty — Percutaneous BAV is performed according to the standard retrograde technique. The measurement of the trans-aortic gradient is given by two catheters placed one in the left ventricle, the other in ascending aorta. An extra stiff wire is placed in the left ventricular cavity. A balloon (size fitting the valve annulus) is inserted over the wire and a series of three inflations is performed at nominal pressure.
  The procedure terminates in case of:
  1. Reduction of the mean aortic gradient ≥50%.
  2. Aortic pressure drop during the inflations, indicative of valve orifice sealing.
  3. Intraprocedural complication.
  4. Poor compliance of the patient. If none is met, the balloon is changed with a bigger one and a new series of three inflations performed. Aortic gradient is finally recorded.

SUMMARY:
Pilot interventional study, without drug, randomized 1: 1, open-label comparison of efficacy and safety between the technique of percutaneous balloon aortic valvuloplasty without rapid ventricular pacing vs valvuloplasty during rapid ventricular pacing (using a temporary pacemaker device with CE mark). It is expected to enroll 100 patients. Randomization is done through a dedicated computer program.

DETAILED DESCRIPTION:
The aim is to compare, in terms of procedural success and safety, the procedure of percutaneous balloon aortic valvuloplasty (BAV) without rapid ventricular pacing with the same procedure carried out with the aid of rapid ventricular pacing.

It is a pilot study with the objective to enroll 100 consecutive patients matching inclusion and exclusion criteria who are randomized 1:1 in two arms: in the first patients undergo procedure of BAV without rapid pacing, in the second BAV with rapid ventricular pacing able to help in balloon stabilization during inflations.

Efficacy will be studied analysing changes in transvalvular gradient from baseline to post-BAV. Safety outcomes will be collected both at discharge and at 30-day. Other procedural data will be object of direct comparison.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of severe symptomatic aortic valve stenosis.
* no immediate indication to aortic valve replacement (AVR).
* indication to balloon aortic valvuloplasty (BAV).
* written expression of informed consent.

Exclusion Criteria:

* clinical presentation in cardiogenic shock at the time of BAV.
* clinical presentation in acute pulmonary edema not previously stabilized by medical therapy.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-04; Primary Completion 2015-12 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy endpoint: trans-aortic gradient reduction ≥ 50% measured with echocardiography from baseline to post BAV (analysis intention to treat). | Post-procedural, on average 30 minutes after the procedure.
  Echocardiography performed 30 minutes after the procedure.
Composite safety endpoint: death, myocardial infarction, stroke, acute aortic valve insufficiency, major bleeding (BARC classification ≥3) | 30-day

SECONDARY OUTCOMES:
Trans-aortic gradient reduction ≥ 50% measured with echocardiography from baseline to post BAV (analysis per treatment). | Post-procedural, on average 30 minutes after the procedure.
  Echocardiography performed 30 minutes after the procedure.
Trans-aortic gradient reduction from 30 to 49% | Post-procedural, on average 30 minutes after the procedure.
  Echocardiography performed 30 minutes after the procedure.
Haemodynamic trans-aortic gradient reduction ≥ 50% | Just after last balloon inflation, on average 3 minutes after BAV
Haemodynamic trans-aortic gradient reduction from 30 to 49% | Just after last balloon inflation, on average 3 minutes after BAV
Overall mortality | 30-day
Cardiovascular mortality | 30-day
Ictus incidence | 30-day
Acute myocardial infarction | 30-day
Acute severe aortic insufficiency | Just after last balloon inflation, on average few seconds after BAV
Major bleeding (BARC ≥3) | 30-day
New cardiovascular hospital admission | 30-day
Evaluation of variations of the aortic valve area, and the maximum and averageaortic gradient by echocardiography from pre to post procedure | Post-procedural, on average 30 minutes after the procedure.

OTHER OUTCOMES:
Compare change in transvalvular gradient pre and post BAV measured between the left ventricle and aorta (LV-Ao) vs gradient measured between the left ventricle and femoral artery (LV-periphery). | Just after last balloon inflation, on average 3 minutes after BAV
Acute kidney injury | at hospital discharge, on average 3 days after BAV
Hospitalization duration | at hospital discharge, on average 3 days after BAV

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Marzocchi, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- Institute of Cardiology, Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy